CLINICAL TRIAL: NCT02113631
Title: Comparative Effectiveness and Tolerability of Boceprevir vs Telaprevir and Re-assessment of Treatment Duration in Patients With Chronic Hepatitis C
Brief Title: Comparative Effectiveness and Tolerability of Boceprevir vs Telaprevir
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yngve Falck-Ytter, MD, Louis Stokes VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #: 11064-H40
Record Dates: First submitted 2014-03-30; First posted 2014-04-14 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic; Cirrhosis
Keywords: Hepatitis C treatment,; Boceprevir,; Telaprevir,; Safety; Effectiveness; Head-to-head trial
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis | interventions — telaprevir; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telaprevir (Active Comparator): Telapravir was administer with Peg-IFN and Ribavirin as per package insert Dose Telaprevir : PO, tablet 1125 mg BID for 12 weeks
  Interventions: Drug: Telaprevir; Drug: Peg-IFN; Drug: Ribavirin
- Boceprevir (Active Comparator): Boceprevir was administer with Peg-IFN and Ribavirin as per package insert Dose Boceprevir PO capsule, 800mg TID for up to 44 weeks
  Interventions: Drug: Boceprevir; Drug: Peg-IFN; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir
  Other Names: INCIVEK
  Arms: Telaprevir
Drug: Boceprevir
  Other Names: Victrelis
  Arms: Boceprevir
Drug: Peg-IFN — Administration 45-180mcg in 0.5 ml solution s.c. weekly for 24-48 weeks
  Other Names: Peg-Interferon alfa-2a, Pegasys
Drug: Ribavirin — Administration: 200 mg capsules; 800 mg-1200 mg daily for 24-48 weeks
  Other Names: Copegus

SUMMARY:
1. The primary objective is to study the comparative effectiveness and tolerability of boceprevir vs. telaprevir in HCV treatment, within the VA population.
2. The secondary objective:

   * Resource use: recording of differences in resource use, such as direct costs (e.g., drug acquisition costs) and other indirect cost (e.g., staff utilization etc.) as the study will not only derive data by comparing those two drugs but also study the effect on different treatment lengths.

DETAILED DESCRIPTION:
This is a randomized clinical trial comparing the effectiveness and safety of boceprevir and telaprevir.

Recruitment of current eligible subjects will occur during their regular appointments at the Hepatitis C clinic. Eligible patients will have already been cleared for Hepatitis C treatment through their screening period which is including blood work, liver biopsy, urine collection/analysis, pregnancy screening and behavioral/mental health screening. On one of their standard visits to the Hepatitis C clinic, the health care provider(who is also research staff) or research staff will provide a consent form that the patient may take home and read more about the study.

On the day of enrollment, which will also be the first day of treatment, health care providers within the Hepatitis C clinic will describe the study to the patient or refer them to one of the research for completion of these tasks. The consent form will be explained in detail at this meeting, and the patient will have the opportunity to ask questions and make comments about the study.

Study subjects will initially be stratified into 6 groups (1a. treatment naives without cirrhosis and b. with compensated cirrhosis ; 2a. prior treatment experienced non-responders without cirrhosis and b. with cirrhosis; 3a. prior treatment experienced relapsers without cirrhosis and b. with cirrhosis). Patients in each of these groups will be randomized using random number table and allocation concealment will be achieved by using serially numbered, opaque, sealed envelopes into one of two study groups. The first group will receive boceprevir with Peg-IFN and ribavirin as indicated by package insert, and the second group will receive telaprevir with Peg-IFN and ribavirin as indicated by its package insert. All other stratified groups will receive protease inhibitor therapy as indicated by the FDA product labeling.

Safety and effectiveness assessments will be conducted at study entry, PI therapy week 0, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 42 and 48, if applicable. Those are SOC visits during the treatment period and they will include blood tests, complete review of systems, and physical exams. Patients in all groups will be assessed for sustained viral response (SVR) at 12 and 24 weeks after the last dose of the medication is administered.

Identical to SOC, safety and effectiveness assessments will be determine by health care providers and the adjudication committee, the latter of which will be unaware of the treatment arm of the patients. Members of the adjudication committee will be independent of the treating clinicians, and will be responsible for adjudicating the following outcomes:

* Viral response
* Adverse effects
* Decision regarding treatment discontinuation, based on adverse effect or virological failure

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Have HCV genotype 1 infection and evidence of chronic hepatitis, as confirmed by a liver biopsy completed within three years prior to enrollment in the study, patients with cirrhosis will not need to undergo biopsy. Patients with compensated liver cirrhosis will be eligible. Patients who have previously been treated under standard of care (Peg-IFN, Ribavrin) and were non-responders, partial responders, or relapsers will also be eligible.
3. Platelet count >60,000/mm3
4. Absolute neutrophil count > 1000/mm3
5. Hemoglobin >11.0 g/dL for females or >12.0 g/dL for males
6. Serum creatinine </=1.5 mg/dL
7. Adequately controlled DM
8. Normal or adequately controlled TSH on prescription medication
9. All other clinical laboratory values within normal limits, unless judged not clinically significant by the investigator
10. Sterile or infertile (defined as vasectomy, tubal ligation, postmenopausal, or hysterectomy), or willing to use an approved method of double-barrier contraception (hormonal plus barrier or barrier plus barrier, eg, diaphragm plus condom) from the time of first dose administration until 6 months after the last dose
11. Capable of understanding instructions, adhering to study schedules and requirements, and willing to provided informed consent

Exclusion Criteria:

1. Positive HIV or HbsAg serology
2. Severe psychiatric or neuropsychiatric disorders including, but not limited to uncontrolled severe depression, history of suicidal ideations or suicide attempt(s), as determinate by SOC psychological evaluation 3 History or clinical manifestations of significant metabolic, hematological, pulmonary, ischemic or unstable heart disease, gastrointestinal, neurological, renal, urological, endocrine, ophthalmologic (including severe retinopathy), or immune mediated disease

4. Chronic hepatic diseases other than hepatitis C 5. Organ or bone marrow transplant 6. Chronic (greater than 30 days) use of immunosuppressive medications including steroids in doses equivalent to 10 mg of prednisone or higher, 30 days prior to and anytime during the course of the study 7. Female patients who are breast-feeding or have a positive pregnancy test at any time during the study 8. Males whose female partners are pregnant 9. Patients who have had a malignancy diagnosed and/or treated within the past 3 years, except for localized squamous or basal cell cancers treated by local excision 10. Patients who have participated in a clinical trial and have received an investigational drug within 30 days prior to screening 11. Current alcoholism or drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety/Adverse Event Outcome Measure | Up to 3 weeks
  Number of Participants with Serious and Non-Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yngve Falck-Ytter, MD, Principal Investigator — Louis Stokes Cleveland VA medical center
Locations (1):
- Louis Stokes Cleveland VA medical center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Flamm SL, Lawitz E, Jacobson I, Bourliere M, Hezode C, Vierling JM, Bacon BR, Niederau C, Sherman M, Goteti V, Sings HL, Barnard RO, Howe JA, Pedicone LD, Burroughs MH, Brass CA, Albrecht JK, Poordad F. Boceprevir with peginterferon alfa-2a-ribavirin is effective for previously treated chronic hepatitis C genotype 1 infection. Clin Gastroenterol Hepatol. 2013 Jan;11(1):81-87.e4; quiz e5. doi: 10.1016/j.cgh.2012.10.006. Epub 2012 Oct 10. PMID 23064222
- [Background] Vierling JM, Davis M, Flamm S, Gordon SC, Lawitz E, Yoshida EM, Galati J, Luketic V, McCone J, Jacobson I, Marcellin P, Muir AJ, Poordad F, Pedicone LD, Albrecht J, Brass C, Howe AY, Colvard LY, Helmond FA, Deng W, Treitel M, Wahl J, Bronowicki JP. Boceprevir for chronic HCV genotype 1 infection in patients with prior treatment failure to peginterferon/ribavirin, including prior null response. J Hepatol. 2014 Apr;60(4):748-56. doi: 10.1016/j.jhep.2013.12.013. Epub 2013 Dec 19. PMID 24362076
- [Background] Bacon BR, Gordon SC, Lawitz E, Marcellin P, Vierling JM, Zeuzem S, Poordad F, Goodman ZD, Sings HL, Boparai N, Burroughs M, Brass CA, Albrecht JK, Esteban R; HCV RESPOND-2 Investigators. Boceprevir for previously treated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1207-17. doi: 10.1056/NEJMoa1009482. PMID 21449784
- [Background] Poordad F, McCone J Jr, Bacon BR, Bruno S, Manns MP, Sulkowski MS, Jacobson IM, Reddy KR, Goodman ZD, Boparai N, DiNubile MJ, Sniukiene V, Brass CA, Albrecht JK, Bronowicki JP; SPRINT-2 Investigators. Boceprevir for untreated chronic HCV genotype 1 infection. N Engl J Med. 2011 Mar 31;364(13):1195-206. doi: 10.1056/NEJMoa1010494. PMID 21449783
- [Background] Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, Marcellin P, Muir AJ, Ferenci P, Flisiak R, George J, Rizzetto M, Shouval D, Sola R, Terg RA, Yoshida EM, Adda N, Bengtsson L, Sankoh AJ, Kieffer TL, George S, Kauffman RS, Zeuzem S; ADVANCE Study Team. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med. 2011 Jun 23;364(25):2405-16. doi: 10.1056/NEJMoa1012912. PMID 21696307
- [Background] Zeuzem S, Andreone P, Pol S, Lawitz E, Diago M, Roberts S, Focaccia R, Younossi Z, Foster GR, Horban A, Ferenci P, Nevens F, Mullhaupt B, Pockros P, Terg R, Shouval D, van Hoek B, Weiland O, Van Heeswijk R, De Meyer S, Luo D, Boogaerts G, Polo R, Picchio G, Beumont M; REALIZE Study Team. Telaprevir for retreatment of HCV infection. N Engl J Med. 2011 Jun 23;364(25):2417-28. doi: 10.1056/NEJMoa1013086. PMID 21696308
- [Background] Sherman KE, Flamm SL, Afdhal NH, Nelson DR, Sulkowski MS, Everson GT, Fried MW, Adler M, Reesink HW, Martin M, Sankoh AJ, Adda N, Kauffman RS, George S, Wright CI, Poordad F; ILLUMINATE Study Team. Response-guided telaprevir combination treatment for hepatitis C virus infection. N Engl J Med. 2011 Sep 15;365(11):1014-24. doi: 10.1056/NEJMoa1014463. PMID 21916639
- [Derived] Davitkov P, Chandar AK, Hirsch A, Compan A, Silveira MG, Anthony DD, Smith S, Gideon C, Bonomo RA, Falck-Ytter Y. Treatment Selection Choices Should Not Be Based on Benefits or Costs Alone: A Head-to-Head Randomized Controlled Trial of Antiviral Drugs for Hepatitis C. PLoS One. 2016 Oct 14;11(10):e0163945. doi: 10.1371/journal.pone.0163945. eCollection 2016. PMID 27741230